CLINICAL TRIAL: NCT01054833
Title: A Clinical Evaluation of the Needleless® Sling for the Treatment of Female Stress Urinary Incontinence
Brief Title: Clinical Evaluation of the Needleless® Sling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, KYU-SUNG LEE, Professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-11-019
Record Dates: First submitted 2010-01-20; First posted 2010-01-22 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2013-05

CONDITIONS: Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Needleless sling (Experimental): Needleless® sling
  Interventions: Procedure: Needleless mid-urethral sling

INTERVENTIONS:
Procedure: Needleless mid-urethral sling — The Needleless® sling is intended for use in women as a tension free, sub-urethral slings for the treatment of SUI resulting from urethral hypermobility and/or intrinsic sphincter deficiency. The Needleless sling is a macroporous, monofilament, knitted polypropylene featuring 'Pocket Positioning Anchors' which allow sling placement without needle introducers; thus eliminating a complicated aspect of the surgery (TVT/TOT) and reducing the potential for bladder injury or inguinal pain that can occur during transobturator needle passage. The Needleless sling was approved by KFDA, and now is available in worldwide including Korea.

SUMMARY:
Urinary incontinence which is a major health issue in women affects 30-40% of older women.

Surgical treatments for SUI have undergone many modifications in the last century.

The Needleless Sling System is a one incision, minimally invasive, surgical procedure that has had great acceptance in Europe and has recently received FDA Clearance for use in the United States.

We will evaluate effectiveness and patient reported outcomes for Needleless® sling system (Neomedic International).

This is a prospective, multicenter, registry. Up to 150 women will be enrolled from up to 3 registry sites.

Patients will be evaluated at baseline, peri-operatively, and post-operatively up to 2 months, up to 6 months and at 12 months.

Effectiveness evaluations will include a standing stress test (objective cure), SANDVIK questions (subjective cure) & I-QOL (quality of life measure).

Other evaluations will include type of anesthesia, concurrent surgery, operative time, post-operative pain, length of hospital stay, returning to usual activities, change of lower urinary tract symptoms (BFLUTSSF, voiding diaries), goal achievement and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

A patient must satisfy the following criteria before entering the study:

1. Patient has objective demonstrable signs of stress urinary incontinence (SUI), including patients with ISD. Objective testing includes: standing stress test, urodynamics evaluation, or pad test.
2. Patient is age 18 or older.
3. Patient had a hysterectomy, tubal ligation or is otherwise incapable of pregnancy, or had a negative pregnancy test prior to study entry and has decided to cease childbearing.
4. Patient agrees to participate in the study, including completion of all study-related procedures and evaluations, and documents this agreement by signing the IRB/EC-approved informed consent.

Exclusion Criteria:

* A patient who meets any of the following criteria will be excluded from participating in the study:

  1. Patient has an associated or suspected neurological disease.
  2. Patient is on anti-coagulation therapy.
  3. Patient has received an investigational drug or device in the past 60 days.
  4. Patient has an active lesion or present injury to perineum or urethra.
  5. Patient has a urethral obstruction.
  6. Patient has a significant cystocele > ICS Stage 2.
  7. The subject has active infection upon urine dipstick analysis, defined as ≥ +1 leukocytes or ≥ +1 nitrates (Must reschedule appointment after UTI resolves.)
  8. Patients with combined POP surgery.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-01; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
The result of standing cough stress test at 12 months. | 12 months after the Needleless sling operation

SECONDARY OUTCOMES:
Sandvik Index Questionnaire | 2, 6, 12 months after the Needleless sling operation
Subjective symptom assessment by visual analogue scale | 2, 6, 12 months after the Needleless sling operation
Post-Operative Pain Assessment | postop, 2 months after the Needleless sling operation
Return to Usual Activities Questionnaire | 2 months after the Needleless sling operation
Standing Cough Stress Test | 6, 12 months after the Needleless sling operation
Incontinence Quality of Life Questionnaires (I-QOL) | 6, 12 months after the Needleless sling operation
BFLUTS-SF questionnaire | 6, 12 months after the Needleless sling operation
Patient Satisfaction Questionnaire | 12 months after the Needleless sling operation

CONTACTS AND LOCATIONS:
Overall Officials: Kyu-Sung Lee, Ph.D, Principal Investigator — Samsung Medical Center
Locations (3):
- South Korea (3):
  - Asan Medical center, Ulsan College of Medicine, Seoul
  - Cheil General Hospital & Women's Healthcare Center, College of Medicine, Kwandong University, Seoul
  - Samsung Medical Center, Seoul

REFERENCES:
- [Derived] Carter E, Johnson EE, Still M, Al-Assaf AS, Bryant A, Aluko P, Jeffery ST, Nambiar A. Single-incision sling operations for urinary incontinence in women. Cochrane Database Syst Rev. 2023 Oct 27;10(10):CD008709. doi: 10.1002/14651858.CD008709.pub4. PMID 37888839